CLINICAL TRIAL: NCT00966667
Title: Health Behaviors Among Individuals Diagnosed With Colorectal Cancer
Brief Title: Health Behaviors in Patients Who Have Finished Treatment for Stage I, Stage II, or Stage III Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 130901; R21CA131611 (NIH); P30CA072720 (NIH); K07CA133100 (NIH); CDR0000653167 (Other: NIH); 0220090178 (Other: IRB)
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer
Keywords: cancer survivor; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cancer survivor: cancer survivor

SUMMARY:
RATIONALE: Gathering information over time from patients who have finished treatment for colorectal cancer may help doctors predict which cancer survivors will improve their physical activity and diet.

PURPOSE: This clinical trial is studying health behaviors in patients who have finished treatment for stage I, stage II, or stage III colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To characterize patterns and identify predictors of post-treatment physical activity and dietary changes made by colorectal cancer survivors.

Secondary

* To identify the affective and cognitive effects of post-treatment physical activity and dietary changes in these patients.
* To identify these patients' preferences regarding diet and physical activity health promotion programs.

OUTLINE: This is a multicenter study.

Patients complete surveys at baseline and at 3 and 6 months. A randomly selected subset of 84 patients also receive an activity monitor to be use at each of the 3 time points. The acceptability of their use is assessed and whether activity levels change across the 3 time points and the extent to which they are convergent with self-reported physical activity are examined.

During each survey, questionnaires are administered to assess the following areas: physical/medical characteristics (self-reported), self-efficacy for physical activity, fruit and vegetable consumption, and dietary fat intake; outcome expectations for physical activity, fruit and vegetable consumption, and dietary fat intake; physical activity and diet behavioral self-regulation; illness representations (causal attributions and controllability of recurrence); perceived risk of colorectal cancer (CRC) recurrence; emotional representations of CRC (cancer-related anxiety and worry about cancer recurrence); healthcare provider recommendations to alter physical activity and dietary intake; social influence from important others; current physical activity and dietary intake; and diet and physical activity program preferences. Patients who received the activity monitor are asked feedback on acceptability of them.

Measures of sociodemographics and disease/treatment characteristics (via medical chart review) are recorded.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized or regional colorectal cancer

  * Stage I, II, or III disease
  * Completed treatment within the past 6 weeks
* No previous diagnosis of colorectal cancer

PATIENT CHARACTERISTICS:

* English speaking
* No current evidence of neoplastic disease except for nonmelanoma skin cancer
* No evidence of severe cognitive impairment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer
Sampling Method: Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2009-11; Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Self-efficacy for changing physical activity and dietary practices | 3 yrs
Outcome expectations with regard to physical activity and dietary practices | 3 yrs
Behavioral self-regulation of physical activity and dietary practices | 3 yrs
Perceived role of physical activity and dietary factors in causing colorectal cancer (CRC) and preventing recurrence (CRC illness representations) | 3 yrs
Perceived risk of CRC recurrence | 3 yrs
Cancer-related anxiety and worry about cancer recurrence (emotional representations of CRC) | 3 yrs
Receipt of healthcare provider recommendations to alter physical activity and diet | 3 yrs
Normative influences of family and friends | 3 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Coups, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (14):
- United States (14):
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - JFK Medical Center in Edison, Edison, New Jersey
  - Centrastate Healthcare System, Freehold, New Jersey
  - Robert Wood Johnson University Hospital at Hamilton, Hamilton, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Saint Peters University Hospital, New Brunswick, New Jersey
  - University Medical Center at Princeton, Princeton, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas